CLINICAL TRIAL: NCT02577367
Title: The Effect of Holding Tube Feeding When Administering Levothyroxine on the Mean Percentage of Levothyroxine Dosage Increase in Patients With Hypothyroidism Started on Enteral Feeding
Brief Title: Mean Percentage of Levothyroxine Dosage Increase in Patients With Hypothyroidism Started on Enteral Feeding
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lost interest in current study
Sponsor: Jocelyne Karam (Other)
Collaborators: Maimonides Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jocelyne Karam, Director, Division of Endocrinology, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-05-02
Record Dates: First submitted 2015-09-14; First posted 2015-10-16 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Tube Feeding
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levothyroxine on empty stomach (Experimental): Levothyroxine will be given on empty stomach, by holding enteral feeding for 2 hours before and 2 hours after Levothyroxine administration
  Interventions: Drug: Levothyroxine
- Levothyroxine during feeding (Active Comparator): Levothyroxine will be given while the enteral feeding is running
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — Administer Levothyroxine
  Other Names: Synthroid

SUMMARY:
The study aims to describe the changes in Levothyroxine dosage requirements in patients with hypothyroidism started on enteral feeding, and assess whether giving levothyroxine on empty stomach affects the mean percentage increase expected in Levothyroxine dosage in these patients.

DETAILED DESCRIPTION:
The study will be a Randomized Controlled trial comparing the mean percentage of Levothyroxine dosage change in hypothyroid patients after the starting of enteral feeding in an inpatient setting in two different groups: a control group where Levothyroxine will be administered with continuous enteral nutrition, and an intervention group where enteral nutrition will be held for two hours before and two hours after the Levothyroxine administration.

The enrollment of eligible patients will be over two to three years and follow up will continue for the duration of the hospital stay or 12 weeks, which ever occurs earlier. Eligible patients will have thyroid function tests at enrollment (within three days of the starting of the tube feeding) and afterwards weekly. Levothyroxine dosage will be adjusted by the endocrinology research team according to the thyroid function results. Initial Levothyroxine dosage and subsequent dosages will be recorded and the mean percentage decrease or increase of Levothyroxine dosage required will be measured in each group. An eventual difference between the two groups mean percentage change will be tested for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to Maimonides Medical Center
* Started on Enteral feeding within 3 days of enrollment: tube feeding, Percutaneous Endoscopic Gastrostomy or PEG tube feeding, or Jejunostomy tube feeding.
* History of Hypothyroidism on a stable dose of Levothyroxine for at least four weeks prior to enteral feeding
* TSH 0.2-10 mIU/ml at enrollment

Exclusion Criteria:

* Concomitant administration of medications that affect thyroid function test including Cholestyramine, Sucralfate, Amiodarone, Lithium, Dopamine, Dobutamine and Dilantin at enrollment.
* Pregnancy
* Known untreated disease or surgery of the small intestine specifically the Jejenum.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Mean percentage change of Levothyroxine dosage | 12 weeks
  The Primary outcome will be the measurement of the mean percentage change of levothyroxine dosage ( end of the enrollment dose as compared to baseline dose) in each of the two comparative groups: The control group of patients receiving Levothyroxine during the tube feeding, and the intervention group of patients receiving Levothyroxine on empty stomach (two hours before and two hours after holding the feeding)

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Karam, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No